CLINICAL TRIAL: NCT03502330
Title: A Phase I/Ib Study of APX005M in Combination With Nivolumab and Cabiralizumab in Patients With Advanced Melanoma, Non-small Cell Lung Cancer or Renal Cell Carcinoma Whose Disease Has Progressed on Anti-PD- 1/PD-L1 Therapy
Brief Title: APX005M With Nivolumab and Cabiralizumab in Advanced Melanoma, Non-small Cell Lung Cancer or Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Apexigen America, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000021757; 5P50CA121974-15 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-18 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Advanced Melanoma; Non-small Cell Lung Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — sotigalimab; cabiralizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 Advanced Solid Tumors (Experimental): Cabiralizumab 4mg/kg plus APX005M 0.03 mg/kg administered in 14 day cycles.
  Interventions: Drug: APX005M; Drug: Cabiralizumab
- Cohort 2 Advanced Solid Tumors (Experimental): Nivolumab 240 mg plus Cabiralizumab 4mg/kg plus APX005M 0.03 mg/kg administered in 14 day cycles.
  Interventions: Drug: APX005M; Drug: Cabiralizumab; Drug: Nivolumab
- Cohort 3 Advanced Solid Tumors (Experimental): Cabiralizumab 4mg/kg plus APX005M 0.1 mg/kg administered in 14 day cycles.
  Interventions: Drug: APX005M; Drug: Cabiralizumab
- Cohort 4 Advanced Solid Tumors (Experimental): Nivolumab 240 mg plus Cabiralizumab 4mg/kg plus APX005M 0.1 mg/kg administered in 14 day cycles.
  Interventions: Drug: APX005M; Drug: Cabiralizumab; Drug: Nivolumab
- Cohort 5 Advanced Solid Tumors (Experimental): Cabiralizumab 4mg/kg plus APX005M 0.3 mg/kg administered in 14 day cycles.
  Interventions: Drug: APX005M; Drug: Cabiralizumab
- Cohort 6 Advanced Solid Tumors (Experimental): Nivolumab 240 mg plus Cabiralizumab 4mg/kg plus APX005M 0.3 mg/kg administered in 14 day cycles.
  Interventions: Drug: APX005M; Drug: Cabiralizumab; Drug: Nivolumab
- Cohort 7 Advanced Melanoma (Experimental): Patients will be treated at the estimated APX005M RP2D in combination with nivolumab 240 mg IV and cabiralizumab 4 mg/kg on day 1 of each 14-day cycle.
  Interventions: Drug: APX005M; Drug: Cabiralizumab; Drug: Nivolumab
- Cohort 8 NSCLC (Experimental): Patients will be treated at the estimated APX005M RP2D in combination with nivolumab 240 mg IV and cabiralizumab 4 mg/kg on day 1 of each 14-day cycle.
  Interventions: Drug: APX005M; Drug: Cabiralizumab
- Cohort 9 RCC (Experimental): Patients will be treated at the estimated APX005M RP2D in combination with nivolumab 240 mg IV and cabiralizumab 4 mg/kg on day 1 of each 14-day cycle.
  Interventions: Drug: APX005M; Drug: Cabiralizumab; Drug: Nivolumab

INTERVENTIONS:
Drug: APX005M — APX005M is a humanized Immunoglobulin G (IgG) 1 agonistic monoclonal antibody that binds cluster of differentiation (CD) 40. APX005M is administered by intravenous infusion.
Drug: Cabiralizumab — Cabiralizumab is a humanized Immunoglobulin G (IgG) 4 monoclonal antibody directed against Colony stimulating factor 1 receptor (CSF1R). Cabiralizumab is administered by intravenous infusion.
Drug: Nivolumab — Nivolumab is a humanized IgG4 monoclonal antibody directed against programmed cell death 1 (PD-1). Nivolumab is administered by intravenous infusion.
  Arms: Cohort 2 Advanced Solid Tumors; Cohort 4 Advanced Solid Tumors; Cohort 6 Advanced Solid Tumors; Cohort 7 Advanced Melanoma; Cohort 9 RCC

SUMMARY:
This trial is a phase 1/1b study to evaluate the safety, efficacy, and tolerability of APX005M in combination with nivolumab and cabiralizumab.

The phase 1 dose escalation portion of the study will enroll patients with advanced solid tumors melanoma, non-small cell lung cancer (NSCLC), and renal cell carcinoma (RCC) in 6 cohorts to determine the recommended phase II dose (RP2D) of APX005M.

The phase 1b dose expansion portion will study the triple drug combination separately in the three disease cohorts: melanoma, NSCLC, and RCC.

ELIGIBILITY:
Inclusion Criteria:

Must have one of the following diagnoses:

Melanoma: Unresectable stage III or stage IV melanoma, irrespective of BRAF status, with histologic or cytologic confirmation.

RCC: Histologic or cytologically documented, locally advanced unresectable or metastatic RCC irrespective of histologic subtype

NSCLC: Histologic or cytologically documented, locally advanced or metastatic (i.e. Stage IIIB not eligible for definitive chemoradiotherapy, stage IV, or recurrent) NSCLC. Patients known to harbor an ALK rearrangement or EGFR mutation known to be sensitive to FDA-approved tyrosine kinase inhibitors (TKI), are only eligible after experiencing disease progression (during or after treatment) or intolerance to an FDA approved ALK TKI or EGFR TKI, respectively. Patients with TKI-treated EGFR mutant NSCLC harboring the secondary EGFR T790M tumor must have received prior osimertinib. Patients with crizotinib-treated ALK rearranged NSCLC must have received a next generation ALK inhibitor.

Additional Inclusion Criteria:

1. Biopsy proven metastatic melanoma, NSCLC or RCC whose disease has progressed on a prior regimen containing a PD-1 or PD-L1 inhibitor, without intervening therapy.
2. At least 1 site of disease must be accessible to provide repeat biopsies for tumor tissue. This site may be a target lesion as long as it will not be made unmeasurable by the biopsy procedure.
3. Age ≥18, able to understand and sign the informed consent form.
4. ECOG performance status < 2.
5. Any number of previous treatments. Other prior systemic therapies must have been administered at least 4 weeks before administration of the study drugs; the exception to this is small molecule inhibitors, which must be stopped at least 2 weeks or after five half-lives of the drug, whichever is shorter, prior to the start of the study drugs.
6. Life expectancy of at least 6 months.
7. A history of previously treated brain metastases is allowed, provided that they are stable for at least 4 weeks.
8. Willingness to undergo mandatory tumor biopsy prior to initiation of therapy and before the fifth cycle.
9. Willingness to provide an archival specimen block, if available, for research.
10. Patients must have normal organ and marrow function (as outlined in Section 3.2.2).
11. Female subject of childbearing potential should have a negative urine or serum pregnancy within 24 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential should be willing to use a highly effective contraception (hormonal or IUD) or be surgically sterile, or abstain from heterosexual activity for a period of at least 5 months after the last dose of study drug. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through at least 7 months after the last dose of study drug.
14. Patients must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per RECIST v1.1 criteria.

    a. Tumor sites situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are not considered measurable unless there has been demonstrated progression in the lesion. Sites for biopsy must be distinct from target lesions used for efficacy assessment.
15. Prior focal radiotherapy is allowed. Radiation to brain, pulmonary or intestinal sites must be completed at least 4 weeks prior to study Day 1. There is no time restriction prior to study Day 1 for patients who have received radiation to bone, soft tissue or other sites. No radiopharmaceuticals (strontium, samarium) within 8 weeks before first dose of study drug administration.
16. Prior surgery that requires general anesthesia must be completed at least 1 week before first dose of study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before first dose of study drug administration and patients should have recovered.

Exclusion Criteria:

1. Untreated brain metastases.
2. A patient who has had prior immune therapy or chemotherapy, within 4 weeks prior to study Day 1, or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent will be excluded. The exception is targeted therapy that must have been completed at least 2 weeks or after 5 half-lives, which ever is shorter, prior to study Day 1. Patients who have had prior ipilimumab must have received their last dose no less than 4 weeks prior to study Day 1.

   1. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   2. Note: Toxicity that has not recovered to ≤ Grade 1 is allowed if it meets the inclusion requirements for laboratory parameters.
3. Has had prior treatment with any other CSF1R inhibitor or CD40 agonist
4. Use of corticosteroids to control immune related adverse events at enrollment will not be allowed, and patients who previously required corticosteroids for symptom control must be off steroids for at least 2 weeks. Low-dose steroid use (≤10 mg of prednisone or equivalent) as corticosteroid replacement therapy for primary or secondary adrenal insufficiency is allowed.
5. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to prior treatments with the exception of clinically insignificant adverse events such as alopecia, clinically insignificant laboratory abnormalities, clinically insignificant rash and Grade 2 neuropathy.
6. History of grade 3-4 neurologic or cardiac toxicity or life-threatening liver toxicity poorly responsive to steroids with prior anti-PD-1/anti-PDL1 monotherapy.
7. Presence of leptomeningeal disease.
8. Has active autoimmune disease unrelated to use of immune checkpoint inhibitors that has required systemic treatment in the past year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Pregnancy or breast feeding. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, cabiralizumab or APX005M, breastfeeding must be discontinued if the mother is enrolled on this trial.
10. Patients may not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
11. Either a concurrent condition (including medical illness, such as active infection requiring treatment with intravenous antibiotics or the presence of laboratory abnormalities) or history of a prior condition that places the patient at unacceptable risk if he/she were treated with the study drug or a medical condition that confounds the ability to interpret data from the study.
12. Concurrent, active malignancies in addition to those being studied.
13. Active (non-infectious) pneumonitis.
14. Has a known Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) acute or chronic infection.
15. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
16. History of myocardial infarction or unstable angina within 3 months prior to Cycle 1, Day 1.
17. Prisoners, or subjects who are under compulsory detention
18. Current or history of clinically significant muscle disorders (e.g., myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels
19. History of anti-drug antibodies, severe allergic, anaphylactic, or other infusion-related reaction to a previous biologic agent
20. Concomitant use of statins while on study. However, a patient using statins for over 3 months prior to study drug administration and in stable status without CK rise may be permitted to enroll
21. Open wounds and active skin infections
22. Uveal melanoma in the Phase Ib dose expansion trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Djureinovic D, Weiss SA, Krykbaeva I, Qu R, Vathiotis I, Moutafi M, Zhang L, Perdigoto AL, Wei W, Anderson G, Damsky W, Hurwitz M, Johnson B, Schoenfeld D, Mahajan A, Hsu F, Miller-Jensen K, Kluger Y, Sznol M, Kaech SM, Bosenberg M, Jilaveanu LB, Kluger HM. A bedside to bench study of anti-PD-1, anti-CD40, and anti-CSF1R indicates that more is not necessarily better. Mol Cancer. 2023 Nov 14;22(1):182. doi: 10.1186/s12943-023-01884-x. PMID 37964379
- [Derived] Weiss SA, Djureinovic D, Jessel S, Krykbaeva I, Zhang L, Jilaveanu L, Ralabate A, Johnson B, Levit NS, Anderson G, Zelterman D, Wei W, Mahajan A, Trifan O, Bosenberg M, Kaech SM, Perry CJ, Damsky W, Gettinger S, Sznol M, Hurwitz M, Kluger HM. A Phase I Study of APX005M and Cabiralizumab with or without Nivolumab in Patients with Melanoma, Kidney Cancer, or Non-Small Cell Lung Cancer Resistant to Anti-PD-1/PD-L1. Clin Cancer Res. 2021 Sep 1;27(17):4757-4767. doi: 10.1158/1078-0432.CCR-21-0903. Epub 2021 Jun 17. PMID 34140403

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 9 RCC: Patients will be treated at the estimated APX005M RP2D in combination with nivolumab 240 mg IV and cabiralizumab 4 mg/kg on day 1 of each 14-day cycle.
  APX005M: APX005M is a humanized Immunoglobulin G (IgG) 1 agonistic monoclonal antibody that binds cluster of differentiation (CD) 40. APX005M is administered by intravenous infusion.
  THIS STUDY ARM/COHORT WAS NEVER ACTIVATED DURING THE STUDY.
  Cabiralizumab: Cabiralizumab is a humanized Immunoglobulin G (IgG) 4 monoclonal antibody directed against Colony stimulating factor 1 receptor (CSF1R). Cabiralizumab is administered by intravenous infusion.
  Nivolumab: Nivolumab is a humanized IgG4 monoclonal antibody directed against programmed cell death 1 (PD-1). Nivolumab is administered by intravenous infusion.
Period: Overall Study
Arm/Group | Cohort 1 Advanced Solid Tumors | Cohort 2 Advanced Solid Tumors | Cohort 3 Advanced Solid Tumors | Cohort 4 Advanced Solid Tumors | Cohort 5 Advanced Solid Tumors | Cohort 6 Advanced Solid Tumors | Cohort 7 Advanced Melanoma | Cohort 8 NSCLC | Cohort 9 RCC
Started | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 5 | 3 | 5 | 1 | 5 | 5 | 6 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Advanced Solid Tumors | Cohort 2 Advanced Solid Tumors | Cohort 3 Advanced Solid Tumors | Cohort 4 Advanced Solid Tumors | Cohort 5 Advanced Solid Tumors | Cohort 6 Advanced Solid Tumors | Cohort 7 Advanced Melanoma | Cohort 8 NSCLC | Total
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8 | 42
Age, Continuous [Median (Full Range); unit: years] | 61 [59 to 66] | 58 [40 to 71] | 69 [69 to 73] | 58 [40 to 63] | 61 [60 to 67] | 61 [44 to 84] | 65.5 [55 to 73] | 60.5 [47 to 67] | 61 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 0 | 0 | 2 | 4 | 2 | 12
  Male | 3 | 4 | 1 | 5 | 3 | 4 | 4 | 6 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 5 | 3 | 5 | 3 | 4 | 6 | 8 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8 | 42
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status is a scale that measures one's level of functioning in terms of ability to care for oneself, daily activity, and physical ability (walking, working, etc.) with a range of 0 to 5. A score of 0 indicates performance without restriction whereas a score of 5 indicates death (a higher score indicates worse functioning).
  Participants
    0 | 3 | 4 | 2 | 5 | 1 | 4 | 6 | 2 | 27
    1 | 0 | 2 | 1 | 0 | 2 | 2 | 2 | 6 | 15
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer Type [Count of Participants; unit: Participants]
  Melanoma | 0 | 2 | 2 | 3 | 0 | 5 | 8 | 0 | 20
  Renal Cell Carcinoma (RCC) | 3 | 4 | 1 | 2 | 2 | 1 | 0 | 0 | 13
  Non-small-cell Lung Cancer (NSCLC) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Measured by Assessing Serious Adverse Events (SAEs)and Adverse Events (AEs)
Description: AEs and SAEs will be examined with (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.03.
Time Frame: From study enrollment up to 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Advanced Solid Tumors | Cohort 2 Advanced Solid Tumors | Cohort 3 Advanced Solid Tumors | Cohort 4 Advanced Solid Tumors | Cohort 5 Advanced Solid Tumors | Cohort 6 Advanced Solid Tumors | Cohort 7 Advanced Melanoma | Cohort 8 NSCLC
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8
Participants
  Experienced any SAE | 1 | 3 | 2 | 2 | 2 | 5 | 3 | 5
  Experienced any AE | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8

2. Primary Outcome: Safety and Tolerability Measured by Eastern Cooperative Oncology Group(ECOG) Performance Status
Description: This 5-point scale ranges from full functioning (0) to dead (5)
Time Frame: From study enrollment up to 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Advanced Solid Tumors | Cohort 2 Advanced Solid Tumors | Cohort 3 Advanced Solid Tumors | Cohort 4 Advanced Solid Tumors | Cohort 5 Advanced Solid Tumors | Cohort 6 Advanced Solid Tumors | Cohort 7 Advanced Melanoma | Cohort 8 NSCLC
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 3 | 6 | 8 | 8
Participants
  0 | 1 | 4 | 2 | 3 | 1 | 1 | 4 | 0
  1 | 2 | 2 | 1 | 2 | 2 | 5 | 4 | 8

3. Secondary Outcome: Efficacy Measured by Objective Response Rate (ORR)
Description: ORR will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria v. 1.1. The RECIST categories used for the target lesion are complete response (CR), partial response (PR), stable disease (NR/SD), and progressive disease (PD).
Time Frame: Six months.
Population: Only participants that completed at least 1 follow up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Advanced Solid Tumors | Cohort 2 Advanced Solid Tumors | Cohort 3 Advanced Solid Tumors | Cohort 4 Advanced Solid Tumors | Cohort 5 Advanced Solid Tumors | Cohort 6 Advanced Solid Tumors | Cohort 7 Advanced Melanoma | Cohort 8 NSCLC
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 3 | 5 | 8 | 8
Participants
  complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  partial response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  stable disease (SD) | 2 | 0 | 0 | 0 | 1 | 2 | 3 | 2
  progressive disease (PD) | 1 | 6 | 3 | 5 | 2 | 3 | 5 | 6

4. Other Pre Specified Outcome: Pharmacokinetics (PK) of APX005M Assessed by Area Under the Curve (AUC).
Description: This outcome will be assessed by blood collection.
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Pharmacokinetics (PK) of APX005M Assessed by Minimum Blood Plasma Concentration (Cmin).
Description: This outcome will be assessed by blood collection.
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pharmacokinetics (PK) of APX005M Assessed by Clearance (CL).
Description: This outcome will be assessed by blood collection.
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pharmacokinetics (PK) of APX005M Assessed by Volume of Distribution (Vss)
Description: This outcome will be assessed by blood collection.
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pharmacokinetics (PK) of APX005M Assessed by Peak Plasma Concentration (Cmax).
Description: This outcome will be assessed by blood collection.
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Tissue-based Pharmacodynamics (PD) of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by CD8+ T Cells .
Description: This outcome will be assessed with tissue biopsies.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Tissue-based Pharmacodynamics (PD) of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by CD163+ Macrophages .
Description: This outcome will be assessed with tissue biopsies.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Blood-based Pharmacodynamics (PD) of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by Circulating CD163+ Macrophages .
Description: This outcome will be assessed via blood collection.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Blood-based Pharmacodynamics (PD) of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by Circulating CD8+ T Cells.
Description: This outcome will be assessed via blood collection.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Cytokine-based Pharmacodynamic (PD) Biomarkers of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by CD40L Levels.
Description: This outcome will be assessed via blood collection.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Cytokine-based Pharmacodynamic (PD) Biomarkers of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by IL-10 Levels.
Description: This outcome will be assessed via blood collection.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Cytokine-based Pharmacodynamic (PD) Biomarkers of APX005M, in Combination With Nivolumab and Cabiralizumab Assessed by Interferon-gamma Levels .
Description: This outcome will be assessed via blood collection.
Time Frame: Change from baseline to 8 weeks.
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Efficacy Measured by Progression-free Survival (PFS)
Description: PFS will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria v. 1.1.
Time Frame: From study enrollment up to 6 years.
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Efficacy Measured by Overall Survival (OS)
Description: OS will be ascertained by review of the National Death Index, medical records and follow-up phone calls.
Time Frame: From study enrollment up to 6 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Cohort 1 Advanced Solid Tumors | Cohort 2 Advanced Solid Tumors | Cohort 3 Advanced Solid Tumors | Cohort 4 Advanced Solid Tumors | Cohort 5 Advanced Solid Tumors | Cohort 6 Advanced Solid Tumors | Cohort 7 Advanced Melanoma | Cohort 8 NSCLC
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 5/5 | 0/3 | 0/6 | 2/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/6 | 2/3 | 2/5 | 2/3 | 5/6 | 3/8 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 5/5 | 3/3 | 6/6 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Advanced Solid Tumors (N=3) | Cohort 2 Advanced Solid Tumors (N=6) | Cohort 3 Advanced Solid Tumors (N=3) | Cohort 4 Advanced Solid Tumors (N=5) | Cohort 5 Advanced Solid Tumors (N=3) | Cohort 6 Advanced Solid Tumors (N=6) | Cohort 7 Advanced Melanoma (N=8) | Cohort 8 NSCLC (N=8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Advanced Solid Tumors (N=3) | Cohort 2 Advanced Solid Tumors (N=6) | Cohort 3 Advanced Solid Tumors (N=3) | Cohort 4 Advanced Solid Tumors (N=5) | Cohort 5 Advanced Solid Tumors (N=3) | Cohort 6 Advanced Solid Tumors (N=6) | Cohort 7 Advanced Melanoma (N=8) | Cohort 8 NSCLC (N=8)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 6 (24) | 2 (3) | 3 (15) | 3 (11) | 5 (22) | 5 (22) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (8)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 3 (10)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (2) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 6 (12)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 3 (4)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 4 (8)
Edema face (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 2 (2) | 2 (3) | 4 (4) | 2 (2) | 5 (5) | 6 (8) | 7 (17)
Fever (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 5 (6) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (4) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (3)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 2 (2) | 3 (3)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (6) | 3 (10) | 3 (13) | 3 (7) | 6 (22) | 3 (4) | 4 (9)
Alkaline phosphatase increased (Investigations) | 1 (1) | 5 (8) | 1 (1) | 2 (5) | 2 (3) | 4 (8) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 5 (11) | 3 (12) | 5 (24) | 3 (18) | 6 (36) | 3 (9) | 8 (24)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 4 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 3 (15) | 5 (16) | 3 (11) | 5 (17) | 3 (8) | 6 (19) | 1 (2) | 3 (5)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (5) | 3 (3)
GGT increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (5)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (7) | 1 (1) | 1 (3) | 1 (2) | 2 (6) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 2 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03502330/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03502330/ICF_001.pdf